CLINICAL TRIAL: NCT00446251
Title: The Highly Sensitized Patients: Effects of Rituximab and Mycophenolate Mofetil (MMF) On Anti-Human Leukocyte Antigen (HLA) Antibody Levels In Patients Awaiting Cadaveric Renal Transplant.
Brief Title: Effects of Rituximab and Mycophenolate Mofetil (MMF) on Highly Sensitized Patients Awaiting Renal Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Dr. Connie Davis, University of Washington
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25668-A; 04-0927-A 05 (Other: University of Washington HSD study number)
Expanded Access: Available
Record Dates: First submitted 2007-03-09; First posted 2007-03-12 (Estimated); Results first posted 2010-03-29 (Estimated); Last update posted 2010-04-06 (Estimated); Status verified 2010-03

CONDITIONS: Kidney Failure, Chronic; Diabetic Nephropathies; Glomerulonephritis, IGA; Hypertension, Renal
Keywords: Dialysis; Kidney; Renal; Nephropathy; Glomerulonephropathy; Immunosuppression; Graft; Compatibility; Transplant; Diabetes; Hypertension; Transplantation, Kidney
MeSH Terms: conditions — Kidney Failure, Chronic; Diabetic Nephropathies; Glomerulonephritis, IGA; Hypertension, Renal; Kidney Diseases; Diabetes Mellitus; Hypertension | interventions — Rituximab; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Rituximab — Rituximab dose is 1,000 mg given as an IV infusion every two weeks for 2 doses (days 1 and 15).
  Other Names: Rituxan, Rituximab
Drug: Mycophenolate mofetil (MMF) — Cellcept is continued from prior study, taken 500 - 1,000 mg BID, P.O.
  Other Names: mycophenolate mofetil, MMF, Cellcept

SUMMARY:
This is a 12-month phase 2, prospective, open label study to evaluate the effect of rituximab with mycophenolate mofetil (MMF)on the PRA of 14 highly sensitized patients who just completed an 8 month trial of MMF treatment alone. PRA values obtained at study enrollment and at 6 and 12 months on combined therapy as well as the rates of transplant will be compared and evaluated using descriptive analysis.

DETAILED DESCRIPTION:
BACKGROUND: Patients who have been exposed to human tissue by prior transplants, blood transfusion or pregnancy may develop and maintain anti-bodies against these foreign human cells (SENSITIZATION). As a result of sensitization these patients are more likely to reject an organ donated from an individual who possesses a similar human cell marker (ANTIGENIC)profile. These sensitized patients will remain on the kidney transplant waiting list up to twice as long as those who are not pre-sensitized.

The Panel of Reactive Antibodies (PRA) is a test panel used to measure the patient reactivity to human leukocyte cell antigens (HLA). A PRA of 75% means the patient reacted to 75% of the antigens on the panel. A high PRA indicates that the subject already has antibodies and is highly SENSITIZED. Spontaneous decreases in PRA titers rarely occur. Thus the probability of transplantation in sensitized patients is significantly decreased.

RATIONALE for use of Rituximab:

By reducing specific B-cell populations Rituximab is currently used as a treatment in auto-immune diseases such as lupus erythematosus and rheumatoid arthritis and some cancers such as B-cell non-Hodgkin's lymphoma. It has been reported to have a potential roll in decreasing anti-human lymphocyte (HLA) antibodies post transplant. More studies are needed to assess its possible benefit among pre-transplant patients. Vierira et al. ["Rituxan for reduction of anti-HLA antibodies in patients awaiting renal transplantation", Am J Transplantation 2002;2:A870] reported on the use of rituximab in sensitized patients. Nine patients on dialysis with a PRA > 50% were treated with rituximab (n=3 per group) at 50, 150, or 375mg/m2. No significant change was seen in WBC, hemoglobin, platelet count, chemistry, liver enzymes or CMV IgG titers. At three days and 6 months after infusion there was a decline in the B cell count compared to pre-infusion levels. In 44%, a decline in PRA was seen. The patients receiving the higher doses had a larger decrement in antibody titers.

GENENTECH, INC. will provide Rituximab, labeled for investigational use. Rituximab is formulated for IV administration as a sterile product as a sterile, preservative-free liquid concentrate for intravenous (IV) administration.

STUDY DESIGN: This is a 12-month phase 2, prospective, open label study to evaluate the effect of rituximab with mycophenolate mofetil (MMF)on the PRA of 14 highly sensitized patients who just completed an 8 month trial of MMF treatment alone. PRA values obtained at study enrollment and at 6 and 12 months on combined therapy as well as the rates of transplant will be compared and evaluated using descriptive analysis.

Primary Endpoints: The number of subjects who experience a decrement from baseline in their Panel of Reactive Antibody values (PRA I, PRA II) or cPRA (calculated PRA when available) at: baseline, 6 and 12 months of study initiation.

Secondary Endpoints: The number of subjects who received a transplant The number of subjects with a negative crossmatch if transplanted.

STUDY POPULATION: Patients on the kidney transplant waiting list who are currently receiving hemodialysis and who have a Panel of Reactive Antibodies (PRA) titer levels over 50% after completing 8 months of mycophenolate mofetil (MMF) treatment alone.

SCREENING: Subjects will be consented, then screened clinically for occurrence of infection, Tuberculosis exposure and for protective antibodies in response to prior vaccination.

RITUXIMAB DOSAGE AND ADMINISTRATION: The Rituximab dose is 1000mg (1gm) given as a single I.V. infusion for 2 doses (days 1 and 15). No extra dosing will be given. Rituximab may be administered in an outpatient setting. Hypersensitivity reactions may occur. Premedication, consisting of acetaminophen (1gm) and diphenhydramine (50mg or equivalent dose) by mouth 30 to 60 minutes prior to the start of an infusion will be considered before each infusion of Rituximab. Rituximab will not be re-administered after initial dose regimen.

(MMF) Mycophenolate mofetil DOSAGE AND ADMINISTRATION: Dosing of MMF will continue at the highest tolerated dose the subject was taking at the completion of the parent study: "Highly Sensitized Patients: effects of mycophenolate mofetil (MMF) on anti- human lymphocyte antibody (HLA) levels in patients awaiting renal transplant". The dose will be adjusted according to standard practices, gastrointestinal tolerance and WBC count.

CLINICAL AND LABORATORY SAFETY EVALUATIONS:

SCREENING:

* Medical history and documentation of the rationale for treatment of the patient's disease with Rituximab.
* Pregnancy test (serum or urine) for women of childbearing potential must be done prior to initial Rituximab treatment date.
* Medical history to include: age, sex, prior transplant history, blood transfusion history, prior pregnancy history, history of autoimmune disease, infection history over the last 5 years, and immunization history.
* Physical examination, including vital signs, and performance status.
* Hematology (within 2 weeks of treatment): complete blood count (CBC) with differential and platelet count.
* Serum Chemistries: glucose, blood urea nitrogen, serum creatinine, uric acid, total bilirubin, alkaline phosphatase, low density lipoprotein, high density lipoprotein, total protein, albumin, aspartate aminotransferase(AST), alanine aminotransferase (ALT), and serum calcium.
* Serology Testing as appropriate: Hepatitis B, Hepatitis C, HIV
* IgG and IgM total antibody counts.
* Drug Monitoring: Baseline = pre-infusion. Serum drug levels for Ritux will also be measured for safety. Human Anti-Rituximab Antibody (HACA)is a test for presence of antibodies against rituximab.
* Lymphocyte Sub Group: A sub-group of type-B lymphocytes called 'CD-19 Cells' are specifically impacted by Rituximab and will be used as a marker of drug efficacy.

ON GOING EVALUATIONS Post -Treatment:

For safety the total IgG and IgM levels will be monitored and IgG supplemented if levels decrease below normal values. Additionally WBC counts that drop below 3.0 will result in changes in the MMF dose. If serious infections occur MMF will be discontinued. Patients will be followed for one year after initial rituximab infusion.

* Hematology: monitor CBC + differential weekly for 1 month then monthly
* Monthly: PRAs will be monitored monthly through the 12th month of the study. The standard PRA value is the sum of anti-bodies produced by 2 main groups of lymphocytes; Class I and Class II. We will have PRA I and PRA II antibody classes reported separately as well as PRA reporting using a calculation (cPRA).
* Quarterly: Serology Testing as appropriate: Hepatitis B, Hepatitis C, HIV, IgG and IgM total antibody counts.
* Monitor Serum Ritux and HACA levels at baseline, 6 months and 9 months.
* Monitor CD19+ B-cells at baseline, weeks 1, 2, 4, months 3, 6, 9 and 12.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18 - 75, inclusive
* Able and willing to give written informed consent and comply with the requirements of the study protocol
* Outpatient status
* Patients with a Panel of Reactive Antibodies (PRA) over 10% after an 8-month trial of MMF monotherapy
* Patients with updated immunizations for tetanus, influenza, hepatitis B, pneumococcus
* Patients with a negative purified protein derivative(PPD ) screen for tuberculosis (TB)within the last 6 months. If subject has a prior history of TB or positive PPD, documentation of adequate treatment is required.
* Women who are of childbearing potential must have a negative serum pregnancy test prior to being enrolled in the study and agree to use a medically acceptable method of contraception throughout the study and for twelve months (1 year) after completion of treatment.
* Men must agree to use an acceptable method of birth control during treatment and for twelve months (1 year) after completion of treatment.
* Liver enzymes ALT and AST less than 2 times the normal limit.

Exclusion Criteria:

* Active infection
* Receipt of live vaccine within 4 weeks prior to first infusion.
* Previous treatment with rituximab (MabThera® / Rituxan®)
* History of multiple recurrent infections defined as more than 3 urinary tract infections, 2 episodes of pneumonia or 3 episodes of otitis/sinusitis in one year, or more than two dialysis line or peritoneal infections within one year.
* Infection with hepatitis C virus (HCV) or hepatitis B virus(HBV) or human immunodeficiency virus (HIV), lack of documentation of treatment of a positive PPD, pregnant or breast-feeding, baseline leukopenia, white blood cell count (WBC) less than 4.0, thrombocytopenia (platelet count less than 100,000/mm) or difficult to treat anemia, a hematocrit chronically less than 32 on intravenous iron and EPO (erythropoietin) therapy, history of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies.
* Concomitant malignancies or previous malignancies within the last five years, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
* History of psychiatric disorder
* Significant cardiac or pulmonary disease (including obstructive pulmonary disease)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-12; Primary Completion 2008-04 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Connie L Davis, MD, Principal Investigator — University of Washington

REFERENCES:
- [Background] Aranda JM Jr, Scornik JC, Normann SJ, Lottenberg R, Schofield RS, Pauly DF, Miles M, Hill JA, Sleasman JW, Skoda-Smith S. Anti-CD20 monoclonal antibody (rituximab) therapy for acute cardiac humoral rejection: a case report. Transplantation. 2002 Mar 27;73(6):907-10. doi: 10.1097/00007890-200203270-00013. PMID 11923690
- [Background] Dafoe DC, Bromberg JS, Grossman RA, Tomaszewski JE, Zmijewski CM, Perloff LJ, Naji A, Asplund MW, Alfrey EJ, Sack M, et al. Renal transplantation despite a positive antiglobulin crossmatch with and without prophylactic OKT3. Transplantation. 1991 Apr;51(4):762-8. doi: 10.1097/00007890-199104000-00005. PMID 2014527
- [Background] Garrett HE Jr, Groshart K, Duvall-Seaman D, Combs D, Suggs R. Treatment of humoral rejection with rituximab. Ann Thorac Surg. 2002 Oct;74(4):1240-2. doi: 10.1016/s0003-4975(02)03824-9. PMID 12400781
- [Background] Gloor JM, Lager DJ, Moore SB, Pineda AA, Fidler ME, Larson TS, Grande JP, Schwab TR, Griffin MD, Prieto M, Nyberg SL, Velosa JA, Textor SC, Platt JL, Stegall MD. ABO-incompatible kidney transplantation using both A2 and non-A2 living donors. Transplantation. 2003 Apr 15;75(7):971-7. doi: 10.1097/01.TP.0000058226.39732.32. PMID 12698082
- [Background] Hack N, Angra S, Friedman E, McKnight T, Cardella CJ. Anti-idiotypic antibodies from highly sensitized patients stimulate B cells to produce anti-HLA antibodies. Transplantation. 2002 Jun 27;73(12):1853-8. doi: 10.1097/00007890-200206270-00001. PMID 12131677
- [Background] Holechek MJ, Hiller JM, Paredes M, Rickard JC, Montgomery RA. Expanding the living organ donor pool: positive crossmatch and ABO incompatible renal transplantation. Nephrol Nurs J. 2003 Apr;30(2):195-204. PMID 12736998
- [Background] Jillella AP, Dainer PM, Kallab AM, Ustun C. Treatment of a patient with end-stage renal disease with Rituximab: pharmacokinetic evaluation suggests Rituximab is not eliminated by hemodialysis. Am J Hematol. 2002 Nov;71(3):219-22. doi: 10.1002/ajh.10213. PMID 12410580
- [Background] Libetta C, Rampino T, Dal Canton A. Polarization of T-helper lymphocytes toward the Th2 phenotype in uremic patients. Am J Kidney Dis. 2001 Aug;38(2):286-95. doi: 10.1053/ajkd.2001.26092. PMID 11479154
- [Background] Maloney DG, Grillo-Lopez AJ, Bodkin DJ, White CA, Liles TM, Royston I, Varns C, Rosenberg J, Levy R. IDEC-C2B8: results of a phase I multiple-dose trial in patients with relapsed non-Hodgkin's lymphoma. J Clin Oncol. 1997 Oct;15(10):3266-74. doi: 10.1200/JCO.1997.15.10.3266. PMID 9336364
- [Background] Miura S, Okazaki H, Satoh T, Amada N, Ohashi Y. Long-term follow-up of living donor renal transplant recipients sensitized after donor specific blood transfusion. Transplant Proc. 2001 Feb-Mar;33(1-2):1221-3. doi: 10.1016/s0041-1345(00)02395-2. No abstract available. PMID 11267267
- [Background] Nitta K, Akiba T, Kawashima A, Kimata N, Miwa N, Nishida E, Uchida K, Honda K, Yumura W, Nihei H. Characterization of TH1/TH2 profile in uremic patients. Nephron. 2002 Jul;91(3):492-5. doi: 10.1159/000064293. PMID 12119483
- [Background] Reff ME, Carner K, Chambers KS, Chinn PC, Leonard JE, Raab R, Newman RA, Hanna N, Anderson DR. Depletion of B cells in vivo by a chimeric mouse human monoclonal antibody to CD20. Blood. 1994 Jan 15;83(2):435-45. PMID 7506951
- [Background] Schweitzer EJ, Wilson JS, Fernandez-Vina M, Fox M, Gutierrez M, Wiland A, Hunter J, Farney A, Philosophe B, Colonna J, Jarrell BE, Bartlett ST. A high panel-reactive antibody rescue protocol for cross-match-positive live donor kidney transplants. Transplantation. 2000 Nov 27;70(10):1531-6. doi: 10.1097/00007890-200011270-00023. PMID 11118102
- [Background] Takeda A, Uchida K, Haba T, Tominaga Y, Katayama A, Kobayashi T, Oikawa T, Morozumi K. Acute humoral rejection of kidney allografts in patients with a positive flow cytometry crossmatch (FCXM). Clin Transplant. 2000;14 Suppl 3:15-20. doi: 10.1034/j.1399-0012.2000.0140s3015.x. PMID 11092347
- [Background] Yokoyama T, Nitta K, Futatsuyama K, Hayashi T, Honda K, Uchida K, Kawashima A, Yumura W, Nihei H. Identification of T helper cell subsets in continuous ambulatory peritoneal dialysis patients. Nephron. 2001 Oct;89(2):215-8. doi: 10.1159/000046070. PMID 11549905
- [Background] Vieira CA, Agarwal A, Book BK, Sidner RA, Bearden CM, Gebel HM, Roggero AL, Fineberg NS, Taber T, Kraus MA, Pescovitz MD. Rituximab for reduction of anti-HLA antibodies in patients awaiting renal transplantation: 1. Safety, pharmacodynamics, and pharmacokinetics. Transplantation. 2004 Feb 27;77(4):542-8. doi: 10.1097/01.tp.0000112934.12622.2b. PMID 15084932

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the parent study: "Highly Sensitized Patients: effects of mycophenolate mofetil (MMF) on anti-human lymphocyte antibody levels in patients awaiting renal transplant" study" at 8 months if the subject had not experienced a 10% or greater reduction in Panel of Reactive Anti-bodies(PRA.
Pre-assignment Details: Single arm study: all subjects received 2 Rituximab infusions of 1,000 mg. Subjects were kept at their highest tolerated dose of mycophenolate mofetil(MMF)from parent study.
Groups:
- Rituximab Infusion and Mycophenolate Mofetil Group: Rituximab was administered by IV infusion at a dose of 1000 mg (1 g) on Days 1 and 15 to subjects already on 8 months of oral mycophenolate mofetil mono therapy (@ 500 - 1,000 mg twice daily as tolerated).
Period: Overall Study
Arm/Group | Rituximab Infusion and Mycophenolate Mofetil Group
Started | 14 (14 subjects were enrolled in this Rituximab-mycophenolic mofetil group.)
Completed | 9
Not Completed | 5
Not completed — On-study Transplants | 2
Not completed — Rituximab Infusion Reaction | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab Infusion and Mycophenolate Mofetil Group
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 41.3 (8.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects Who Experience a Decrease in Their Panel of Reactive Antibodies (PRA) at 6 Months Post Rituximab Infusion.
Description: the number of subjects who experience a decrease in their Panel of Reactive Antibodies (PRA) at 6 months and 12 months post Rituximab infusion
Time Frame: Month 6 from start of study
Population: 12 subjects received the full dose of Rituximab AND continued to month 6 post infusion.
Measure: Number; unit: Participants
Arm/Group | Rituximab Infusion and Mycophenolate Mofetil Group
Number analyzed (Participants) | 12
Participants | 6

2. Secondary Outcome: The Number of Subjects Who Experience a Change From Baseline in Their Panel of Reactive Antibody (PRA) Titers at 12 Months Post Rituximab Infusion.
Time Frame: Month 12 from start of study
Measure: Number; unit: Participants
Arm/Group | Rituximab Infusion and Mycophenolate Mofetil Group
Number analyzed (Participants) | 12
Participants | 6

3. Secondary Outcome: The Number of Subjects With a Negative Crossmatch at the Time of Transplant.
Time Frame: Month 12 from start of study
Population: As per protocol each subject was entered with intention to treat.
Measure: Number; unit: Participants
Arm/Group | Rituximab Infusion and Mycophenolate Mofetil Group
Number analyzed (Participants) | 12
Participants | 0

ADVERSE EVENTS:
Arm/Group | Rituximab Infusion and Mycophenolate Mofetil Group
Serious Adverse Events (participants affected / at risk) | 1/14
Other Adverse Events (participants affected / at risk) | 3/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab Infusion and Mycophenolate Mofetil Group (N=14)
Chest pain (Cardiac disorders) | 1 (1) — Chest pain ensuing after Rituximab infusion in subject with known coronary artery disease.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab Infusion and Mycophenolate Mofetil Group (N=14)
Leukopenia (Immune system disorders) | 1 (1)
Infusion reaction (Immune system disorders) | 2 (2) — Two infusion reactions: shortness of breath and backpain with moderately increased body temp and blood pressure.
Pancreatitis (Gastrointestinal disorders) | 1 (1) — 7 days post infusion the subject developed acute pancreatitis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days